CLINICAL TRIAL: NCT03263585
Title: Identification and Treatment of Back Pain in Elderly Women With Osteoporosis
Brief Title: Treatment With a Spinal Orthosis Compared to Equipment Group Training and a Control Group
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helena Salminen (Other)
Collaborators: Medi GmbH & Co.KG (Unknown)
Responsible Party: Sponsor-Investigator, Helena Salminen, PI, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: dnr 2011/142-31/3
Record Dates: First submitted 2017-06-26; First posted 2017-08-28 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Osteoporosis; Vertebral Fracture; Back Pain; Elderly Women
Keywords: Osteoporosis; Vertebral Fracture; Back Pain; Spinal orthosis; Elderly women
MeSH Terms: conditions — Osteoporosis; Spinal Fractures; Back Pain

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Spinal orthosis group (Active Comparator): Women wearing the spinal orthosis Spinomed for 6 months at least 2 hours a day.
  Interventions: Device: Spinal orthosis Spinomed
- Equipment training group (Active Comparator): Women training once a week in an equipment training group led by a physiotherapist for six months.
  Interventions: Other: Equipment training
- Control (No Intervention): Women in the control group get no intervention for six months.

INTERVENTIONS:
Device: Spinal orthosis Spinomed
  Arms: Spinal orthosis group
Other: Equipment training
  Arms: Equipment training group

SUMMARY:
Background: Back pain and osteoporosis with vertebral fractures are common conditions in elderly women and significantly affect their quality of life. A common complication of osteoporosis are vertebral fractures. Treatment with bone-specific drugs does often not help the pain condition caused by the vertebral fractures even when the progress of the disease has decreased. Vertebral fractures often result in deformation of the spine and poorer quality of life of the individual. The spinal kyphosis also affects the lung function and the effect of the kyphosis itself is severe. Alternative treatments of back pain may lead to reduced drug demand for pain. Physical activity is one of the most important factors that regulates bone mass and can also affect balance and fall risk positively. The back orthosis that we intend to use in the treatment study has been shown in some previous scientific studies to strengthen the muscles in the back and also decrease the pain.

Purpose: The purpose of the study was to evaluate the effect of treatment of back pain in elderly women with an activating functional orthosis versus treatment with a group of physiotherapeutic tools and a control group for a six-month treatment period and follow-up after 12 months from the start of study. The aim was also to study elderly women with osteoporosis and back pain in a follow-up study of a cohort of women at high risk of osteoporotic fractures, with focus on back pain, functional capacity and quality of life.

The aim was to study the effect of treatment with activating functional orthosis versus physiotherapeutic treatment in a group and a control group without treatment. The main outcomes will be the experienced perceived back pain and back extensor strength. Additional outcomes will be quality of life, balance, lung function and kyphosis. Biochemical markers for pain will be measured in the RCT (Randomized Controlled Trial).

Significance: Evaluation of alternative treatment methods such as exercise by a physiotherapist and treatment with a functional orthosis will give new additional treatment options for our patients. An activating functional orthosis could reduce the use of analgesics and increase the quality of life of the affected women.

DETAILED DESCRIPTION:
The aims: 1. Identification in a population-based cohort of elderly women the occurrence of vertebral fractures, back pain and their impact on quality of life.

2. To study the effect of treatment with a functional activating orthotic and physiotherapy in an equipment training group, both in comparison with a control group, on the perceived pain, back extensor muscle strength, quality of life, balance and incidence of falls, lung function and kyphosis.

3. Qualitative study of how participants experienced treatment and exercise in an activating orthotic. The investigators hypothesis was that a functional orthotic could be a complementary treatment method that could reduce the use of analgesics and increase the quality of life.

The purpose of the study was to evaluate the effect of treatment of back pain in elderly women with an activating spinal orthotic versus treatment with a physiotherapy equipment training group and a control group for a six-month treatment period and a follow-up six months after the end of treatment. The aim was also to identify the occurrence of vertebral fractures in a cohort of elderly women and to investigate their perceived quality of life.

Background: Osteoporosis is a condition in the skeleton that is characterized by reduced bone density and an increased risk of fractures [1]. Back pain and osteoporosis with vertebral fractures are common conditions in elderly women that significantly affect their quality of life. Vertebral fractures are the most common type of osteoporotic fracture [2]. Vertebral fractures are underdiagnosed and are a major problem. It is estimated that only one third of vertebral fractures are clinically detected [3]. The lifetime risk for a Swedish postmenopausal woman to get a clinically detected vertebral fracture is approximately 15% [4].

In the acute phase, a vertebral fracture is very painful and in the aftermath the vertebral fracture often leads to chronic back pain, increased kyphosis mainly located to the thoracic and lumbar spine, reduction in body height and impaired lung function. There exists a correlation between increased kyphosis and increased risk of falls [5]. Vertebral fractures can affect important daily activities and provide a lower health-related quality of life [6-8].

Treatment with bone-specific drugs does not relieve the back pain caused by the vertebral fractures despite improvement in the state of the disease. The kyphosis also affects lung function, and the effects of the kyphosis itself have previously been considered as very severe.

An important part in the treatment of patients with osteoporosis is physical therapy with an equipment training group. The goal is to maintain or increase mobility, strength and balance that can improve health-related quality of life and prevent fractures. Training of the back extensor muscles have shown to have a positive impact on health-related quality of life, reduce back pain, and training could also affect fear of falling positively [5, 9].

A German randomized controlled study from 2004 and one from 2011 has shown a positive effect of treatment with an activating spinal orthotic on body posture, back extensor muscular strength and quality of life in elderly women with osteoporosis and vertebral fractures [10, 11]. It was shown that wearing the spinal orthotic, back extensor muscle strength was increased through biofeedback. Training with the spinal orthotic also resulted in a significant decrease of the kyphosis, which also affected lung function and body height positively.

The investigators now intend, in a randomized controlled study, to compare training in an activating spinal orthotic with training in an equipment training group, led by a physiotherapist, to see if positive results can be obtained in reduced back pain, increased muscle strength in back extensor muscle, increasing mobility, and decreased kyphosis in the thoracic and lumbar spine. It can also lead to improved lung capacity, and further increased health-related quality of life. If the training method in the activating spinal orthotic appears to work, it would improve the possibilities to train and treat patients with osteoporosis, vertebral fractures and back pain.

Design A. A cross-sectional study of cohort elderly women regarding the occurrence of vertebral fractures and their impact on health related quality of life and back pain.

B. A randomized controlled study where the effect of treatment with an activating spinal orthotic is compared with training in an equipment training group led by a physiotherapist and with an untreated control group for a six-month treatment period and a follow-up six months after the end of the treatment period.

C. A qualitative study with interviews in focus groups were the participating women may describe their experiences of training in an activating spinal orthotic and how they experience health related quality of life during the treatment period.

Methods Cross-sectional study All 186 women who participated in the follow-up study of the Primos project, a population-based cohort study in Stockholm were invited to participate in the current study [12-15]. All these women have been re-examined clinically in a longitudinal follow-up study with bone density measurements of the hip, lumbar spine, whole body and heel, clinical risk markers for osteoporosis and metabolic disease, nutritional status and a balance tests in 2007-2009.

Women interested in participating in the study got an invitation to a study visit. During the study visit, written and oral information about the study was being given and then the women signed an informed consent.

Examinations in the cross sectional study

1. Clinical examination of the back, assessment of kyphosis, body weight and height, assessment of quality of life with SF-36 (Short Form-36) Health Survey) [16, 17], Qualeffo-41(Quality of life questionnaire of the European Foundation for Osteoporosis) [18, 19, 20] and EQ-5D (EuroQol-5Dimensions) Manual Balance Test, assessment of Back Extensor muscle strength. Evaluation of hand grip strength with a JAMAR hydraulic hand dynamometer.

   Assessment of physical performance and back pain using questionnaires, VAS (Visual Analogue Scale) scale and Borg CR-10 (Categoric Rate). Previous frequency of falls. Use of drugs and analgesics. Examination with spirometry and PEF (Peak Expiratory Flow).
2. Referral to X-ray of the thoracic and lumbar spine for assessment of the occurrence of vertebral fractures.

Randomized controlled trial: The investigators expect to recruit at least 108 women, randomized to three treatment arms with approximately 36 women in each arm.

1. Treatment with the activating spinal orthotic Spinomed (Medi-Bayreuth, Bayreuth Germany), maximum of two hours per day with gradual escalation of the time initially. Adaptation of the spinal orthotic is to be performed by an orthopedic technician.
2. Equipment training group led by a physiotherapist once a week with a special training program tailored to elderly women with osteoporosis and back pain.
3. Control group. Power calculation Primary endpoints in the treatment study are a change in experienced back pain, measured with VAS scale and Borg CR-10.

With a sample size of 99 subjects, I e 33 women in each arm analyzed by ANOVA, 88% power at the alpha 5% level is able to detect if there is a difference between the groups. With a possible anticipated drop-out of about 10% of the participants during the study, the investigators have decided to include 36 women in each group, I e a total of 108 women.

Recruitment

1. Participation is offered to women aged ≥ 60 years from the Primos project.
2. Recruitment through an invitation of women aged ≥ 60 years who participated in osteoporosis school in the last five years at Rehab City Kungsholmen.
3. Recruitment through advertisements in daily newspapers and ads in appropriate web forums (eg website for the National Association of Osteoporotic ROP) Flow chart Baseline

1. Clinical examination of the back, assessment of spinal curvature and of muscle strength of the back extensors, measurement of weight and height, assessment of health related quality of life with SF-36 [16, 17], Qualeffo-41 [18, 19, 20] and EQ-5D [21]. Manual balance test. Evaluation of hand grip strength with JAMAR dynamometer.

Assessment of physical performance and perceived pain using questionnaires, VAS scales and Borg CR-10. Examination with spirometry and PEF. Assessment of previous falls during the last year and other risk factors for osteoporotic fractures. Use of drugs and analgesics.

2. Referral to X-ray of the thoracic and lumbar spine for assessment of the occurrence of vertebral fractures. 3. Blood sample of 20 ml venous blood for analysis of substance P and CGRP (Calcitonin Gene Related Peptide) and IL-6 (Interleukin-6). Storage of samples: frozen in -70gr freezer until analyzes at a special research laboratory where one of the co-worker in the study is responsible for the analyzes.

Collaboration with the same radiological clinic at Karolinska University Hospital Solna for all X-ray examinations.

Follow-up after 1 month Pain drawing, pain measured by VAS-scale and Borg CR-10. For the spinal orthotic group adjustment of the spinal orthotic. Report of falls during last month. Use of drugs and analgesics.

Visit 2 after 3 months Clinical examination: functional assessment of the back, muscle strength of the back extensors, hand grip strength with JAMAR, pain drawing, manual balance test, back pain measured by VAS scale and Borg CR-10, EQ-5D, SF-36, Qualeffo-41. Adjustment of spinal orthotic. Spirometry. Weight and height. Report of falls since visit 1. Use of drugs and analgesics.

Visit 3 after 6 months Clinical examination: Functional assessment of the back. Manual balance test, muscle strength of the back extensors, grip strength with JAMAR, pain drawing, back pain measured by VAS-scale and Borg CR-10, EQ-5D, SF-36, Qualeffo-41. Spirometry. Weight and height. Assessment of spinal curvature. Report of falls since 3 month visit. Use of drugs and analgesics. Blood sample for substance P, IL-6 and CGRP analysis (Calcitonin Gene Related Peptide).

Qualitative group interviews in the Spinomed groups, using a semi-structured interview guide will be performed after the participants have completed their participation in the RCT.

Follow-up 12 months after study start Women in the group treated with the spinal orthotic Spinomed may continue to use the orthotic on their own initiative between 2 hours to a maximum of 4 hours per day, but without follow-up until after six months. Follow-up with reporting falls in a logbook once a week.

Women in the equipment training group receive a home exercise program they can continue at home, but without follow-up until after six months Visit 4 six months after end of treatment Clinical examination: Functional assessment of the back, manual balance test, muscle strength of the back extensors, hand grip strength with JAMAR, pain drawing, back pain measured with VAS scale and Borg CR-10. EQ-5D, Qualeffo-41, SF-36, Spirometry, Weight and height. Falls frequency. Assessment of spinal curvature. Use of drugs and analgesics.

ELIGIBILITY:
Inclusion Criteria

* Woman aged ≥ 60 years
* Osteoporosis according to DXA (Dual X-Ray Absorptiometry) hip (femoral neck or total hip) or lumbar spine.
* Back pain.

Exclusion Criteria

* Diagnosed symptomatic spinal stenosis
* Difficulty to participate in the activities included in the study due to health problems.
* Difficulty to participate in equipment training group.
* Inability to be able to complete wearing the spinal orthosis.
* Language difficulties
* Cognitive difficulties
* Visual problems

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2012-05-03 (Actual); Primary Completion 2012-11-22 (Actual); Study Completion 2014-12-22 (Actual)

PRIMARY OUTCOMES:
Back pain | Baseline and six months
  Measured with Visual Analogue Scale

SECONDARY OUTCOMES:
Back muscle extensor strength | Baseline and six months
  Measured with DigiMax in newton, women press their back against a pad for 6 seconds, three times.
Borg CR-10 | Baseline and six months
  Back pain measured by Borg CR-10
Kyphosis | Baseline and six months
  Measured by flexicurve ruler
Substance P | Baseline and six months
  Biochemical markers
CGRP Calcitonin Gene Related Peptide | Baseline and six months
  Biochemical markers
IL-6 Interleukin | Baseline and six months
  Biochemical markers
Lung function | Baseline and six months
  Spirometry
Balance | Baseline and six months
  Manual balance test
Gait speed | Baseline and six months
  Women walk 2x15 meter as fast as possible
SF-36 | Baseline and six months
  Health related quality of life
QUALEFFO-41 | Baseline and six months
  Health related quality of life
EQ-5D | Baseline and six months
  Health related quality of life
Hand grip strength | Baseline and six months
  Measured by JAMAR Manometer
Height | Baseline and six months
  Measured by stadiometer in cm
Log book | Baseline and six months
  Back pain measured by log book
Paindrawing | Baseline and six months
  Back pain measured by paindrawing
Falls | Baseline and six months
  Self reported falls

CONTACTS AND LOCATIONS:
Overall Officials: Eeva Helena S Salminen, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Rehab City, Stockholm
  - Liljeholmen Academic Health Centre, Stockholm

IPD SHARING:
Plan to Share IPD: No
Individual participant data is available only for the research group and available for other researchers only after new ethical review and in collaboration

REFERENCES:
- [Background] Assessment of fracture risk and its application to screening for postmenopausal osteoporosis. Report of a WHO Study Group. World Health Organ Tech Rep Ser. 1994;843:1-129. No abstract available. PMID 7941614
- [Background] Cauley JA, Hochberg MC, Lui LY, Palermo L, Ensrud KE, Hillier TA, Nevitt MC, Cummings SR. Long-term risk of incident vertebral fractures. JAMA. 2007 Dec 19;298(23):2761-7. doi: 10.1001/jama.298.23.2761. PMID 18165669
- [Background] Delmas PD, van de Langerijt L, Watts NB, Eastell R, Genant H, Grauer A, Cahall DL; IMPACT Study Group. Underdiagnosis of vertebral fractures is a worldwide problem: the IMPACT study. J Bone Miner Res. 2005 Apr;20(4):557-63. doi: 10.1359/JBMR.041214. Epub 2004 Dec 6. PMID 15765173
- [Background] Kanis JA, Johnell O, Oden A, Borgstrom F, Zethraeus N, De Laet C, Jonsson B. The risk and burden of vertebral fractures in Sweden. Osteoporos Int. 2004 Jan;15(1):20-6. doi: 10.1007/s00198-003-1463-7. Epub 2003 Oct 31. PMID 14593450
- [Background] Kasukawa Y, Miyakoshi N, Hongo M, Ishikawa Y, Noguchi H, Kamo K, Sasaki H, Murata K, Shimada Y. Relationships between falls, spinal curvature, spinal mobility and back extensor strength in elderly people. J Bone Miner Metab. 2010;28(1):82-7. doi: 10.1007/s00774-009-0107-1. Epub 2009 Aug 19. PMID 19690799
- [Background] Hallberg I, Bachrach-Lindstrom M, Hammerby S, Toss G, Ek AC. Health-related quality of life after vertebral or hip fracture: a seven-year follow-up study. BMC Musculoskelet Disord. 2009 Nov 3;10:135. doi: 10.1186/1471-2474-10-135. PMID 19886998
- [Background] Papaioannou A, Kennedy CC, Ioannidis G, Brown JP, Pathak A, Hanley DA, Josse RG, Sebaldt RJ, Olszynski WP, Tenenhouse A, Murray TM, Petrie A, Goldsmith CH, Adachi JD. Determinants of health-related quality of life in women with vertebral fractures. Osteoporos Int. 2006;17(3):355-63. doi: 10.1007/s00198-005-2020-3. Epub 2005 Dec 9. PMID 16341623
- [Background] Strom O, Borgstrom F, Zethraeus N, Johnell O, Lidgren L, Ponzer S, Svensson O, Abdon P, Ornstein E, Ceder L, Thorngren KG, Sernbo I, Jonsson B. Long-term cost and effect on quality of life of osteoporosis-related fractures in Sweden. Acta Orthop. 2008 Apr;79(2):269-80. doi: 10.1080/17453670710015094. PMID 18484255
- [Background] Francis RM, Aspray TJ, Hide G, Sutcliffe AM, Wilkinson P. Back pain in osteoporotic vertebral fractures. Osteoporos Int. 2008 Jul;19(7):895-903. doi: 10.1007/s00198-007-0530-x. Epub 2007 Dec 11. PMID 18071648
- [Background] Pfeifer M, Begerow B, Minne HW. Effects of a new spinal orthosis on posture, trunk strength, and quality of life in women with postmenopausal osteoporosis: a randomized trial. Am J Phys Med Rehabil. 2004 Mar;83(3):177-86. doi: 10.1097/01.phm.0000113403.16617.93. PMID 15043351
- [Background] Pfeifer M, Kohlwey L, Begerow B, Minne HW. Effects of two newly developed spinal orthoses on trunk muscle strength, posture, and quality-of-life in women with postmenopausal osteoporosis: a randomized trial. Am J Phys Med Rehabil. 2011 Oct;90(10):805-15. doi: 10.1097/PHM.0b013e31821f6df3. PMID 21681065
- [Background] Salminen H, Saaf M, Ringertz H, Strender LE. Bone mineral density measurement in the calcaneus with DXL: comparison with hip and spine measurements in a cross-sectional study of an elderly female population. Osteoporos Int. 2005 May;16(5):541-51. doi: 10.1007/s00198-004-1719-x. Epub 2004 Sep 21. PMID 15448984
- [Background] Salminen H, Saaf M, Johansson SE, Ringertz H, Strender LE. Nutritional status, as determined by the Mini-Nutritional Assessment, and osteoporosis: a cross-sectional study of an elderly female population. Eur J Clin Nutr. 2006 Apr;60(4):486-93. doi: 10.1038/sj.ejcn.1602341. PMID 16391579
- [Background] Salminen H, Saaf M, Ringertz H, Strender LE. The role of IGF-I and IGFBP-1 status and secondary hyperparathyroidism in relation to osteoporosis in elderly Swedish women. Osteoporos Int. 2008 Feb;19(2):201-9. doi: 10.1007/s00198-007-0463-4. Epub 2007 Sep 14. PMID 17874030
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Lips P, Cooper C, Agnusdei D, Caulin F, Egger P, Johnell O, Kanis JA, Kellingray S, Leplege A, Liberman UA, McCloskey E, Minne H, Reeve J, Reginster JY, Scholz M, Todd C, de Vernejoul MC, Wiklund I. Quality of life in patients with vertebral fractures: validation of the Quality of Life Questionnaire of the European Foundation for Osteoporosis (QUALEFFO). Working Party for Quality of Life of the European Foundation for Osteoporosis. Osteoporos Int. 1999;10(2):150-60. doi: 10.1007/s001980050210. PMID 10501796
- [Background] Lips P, van Schoor NM. Quality of life in patients with osteoporosis. Osteoporos Int. 2005 May;16(5):447-55. doi: 10.1007/s00198-004-1762-7. Epub 2004 Dec 18. PMID 15609073
- [Background] Lips P, Agnusdei D, Caulin F, Cooper C, Johnell O, Kanis J, Liberman U, Minne H, Reeve J, Reginster JY, de Vernejoul MC, Wiklund I. The development of a European questionnaire for quality of life in patients with vertebral osteoporosis. Scand J Rheumatol Suppl. 1996;103:84-5; discussion 86-8. doi: 10.3109/03009749609103757. PMID 8966496
- [Background] Brooks R. EuroQol: the current state of play. Health Policy. 1996 Jul;37(1):53-72. doi: 10.1016/0168-8510(96)00822-6. PMID 10158943
- [Background] Sullivan M, Karlsson J, Ware JE Jr. The Swedish SF-36 Health Survey--I. Evaluation of data quality, scaling assumptions, reliability and construct validity across general populations in Sweden. Soc Sci Med. 1995 Nov;41(10):1349-58. doi: 10.1016/0277-9536(95)00125-q. PMID 8560302
- [Derived] Kaijser Alin C, Uzunel E, Grahn Kronhed AC, Alinaghizadeh H, Salminen H. Effect of treatment on back pain and back extensor strength with a spinal orthosis in older women with osteoporosis: a randomized controlled trial. Arch Osteoporos. 2019 Jan 9;14(1):5. doi: 10.1007/s11657-018-0555-0. PMID 30623268